CLINICAL TRIAL: NCT03815474
Title: Anlotinib Hydrochloride Combined With Epirubicin and Ifosfamide for Locally Recurrent or Metastatic Soft Tissue Sarcoma Patients: a One-arm, Multi-center, Prospective Clinical Trial
Brief Title: Anlotinib Hydrochloride Combined With Epirubicin and Ifosfamide for Soft Tissue Sarcoma Patients
Acronym: ALTER-S005
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Collaborators: First Hospital of China Medical University (Other); Dalian Municipal Central Hospital (Other); The Second Affiliated Hospital of Dalian Medical University (Other); China-Japan Friendship Hospital (Other); The Third Affiliated Hospital of Harbin Medical University (Other); Second Hospital of Jilin University (Other); Daqing Oil Field Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2018012
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2019-07-09 (Actual); Status verified 2019-01

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — anlotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anlotinib & epirubicin& ifosfamide (Experimental): interventions:Anlotinib 12 mg once daily for 14 days tablet by mouth ; epirubicin 30mg/m2 intravenous injection from 1 day to 2 , ifosfamide 1.8g/m2 intravenous injection from 1day to 5day with 6 cycles. Anlotinib 12 mg once daily for 14 days tablet by mouth to progressive disease
  Interventions: Drug: anlotinib

INTERVENTIONS:
Drug: anlotinib — Anlotinib 12 mg once daily for 14 days tablet by mouth ; epirubicin 30mg/m2 intravenous injection from 1 day to 2 , ifosfamide 1.8g/m2 intravenous injection from 1day to 5day with 6 cycles. Anlotinib 12 mg once daily for 14 days tablet by mouth to progressive disease
  Other Names: epirubicin ifosfamide

SUMMARY:
Anlotinib is a multi-target receptor tyrosine kinase inhibitor. It can inhibit the angiogenesis related kinase, such as Vascular Endothelial Growth Factor Receptor (VEGFR), Fibroblast Growth Factor Receptor(FGFR), Platelet-Derived Growth Factor Receptor(PDGFR), and tumor cell proliferation related kinase c-Kit kinase. Anlotinib is an efficient second line therapeutic agent in treatment for metastatic soft tissue sarcoma which has been approved in clinical trials (ALTER-0203).Therefore , this study evaluates the safety and efficacy of anlotinib plus epirubicin and ifosfamide treat the metastatic or advanced soft tissue sarcoma .

DETAILED DESCRIPTION:
This study is planned to be carried out in Liaoning, Jilin and Harbin provinces regional multi-center. 47 cases are preliminarily expected to be included. The study started in January 2019 and ended in December 2019. It is expected that the trial will end in December 2020. This study is a phase 2 study evaluating the safety and efficacy anlotinib and plus epirubicin and ifosfamide treat the metastatic or advanced soft tissue sarcoma .

All those participants need to sign informed consent forms for data collection and use for research purpose before inclusion .Those participants who were not treated with anthracyclines or other tyrosinase inhibitors or angiostatins within the first 6 months should be enrolled.

47 subjects with metastatic or advanced soft tissue sarcoma will receive epirubicin at 30mg/m2/day（day1-2 IV）, ifosfamide at 1.8g/m2/day (day1-5 IV) anlotinib at a dose of 12 mg once daily (day8-21 PO). After 6 treatment cycles,those participants will receive anlotinib at a dose of 12 mg once daily (day8-21 PO) in 21-day cycles until disease progression (defined by RECIST version 1.1) ot unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form prior to patient entry;
* ≥ 18 years of age , regardless of gender；ECOG :0-1;Expected Survival Time: Over 3 months;
* Histologically confirmed diagnosis of un-resectable or recurrent metastatic soft tissue sarcoma, such as: leiomyosarcoma, synovial sarcoma, undifferentiated pleomorphic sarcoma, liposarcoma , angiosarcoma and other sarcomas. The following histologies are excluded: alveolar Soft tissue sarcoma, rhabdomyosarcoma, chondrosarcoma, osteosarcoma, gastrointestinal stromal tumor, humeral cutaneous fibrosarcoma, Ewing sarcoma/primary neuroectodermal tumor, inflammatory myofibroblastic sarcoma and malignant mesothelioma.
* Patients who were not treated with anthracyclines or other tyrosinase inhibitors or angiostatins within the first 6 months should be enrolled.
* Evaluable disease by imaging or physical exam or measurable disease defined as at least one lesion that can be accurately measured according to RECIST version 1.1.
* normal main organs function as defined below: Hemoglobin (Hb) ≥ 80g / L, Neutrophils (ANC) ≥ 1.5 × 109 / L, Platelet count (PLT) ≥ 80 × 109 / L, Serum creatinine (Cr) ≤ 1.5 × normal upper limit (ULN) or creatinine clearance (CCr) ≥ 60ml / min, Blood urea nitrogen (BUN) ≤ 2.5 × normal upper limit (ULN); Total bilirubin (TB) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN; If accompanied by liver metastases, ALT and AST ≤ 5 × ULN Albumin (ALB) ≥ 25 g/L. Doppler ultrasound assessment: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%)
* Women of childbearing potential should agree to use and utilize an adequate method of contraception (such as intrauterine device，contraceptive and condom) throughout treatment and for at least 6 months after study is stopped；the result of serum or urine pregnancy test should be negative within 7 days prior to study enrollment，and the patients required to be non-lactating；Man participants should agree to use and utilize an adequate method of contraception throughout treatment and for at least 6 months after study is stopped.

Exclusion Criteria:

* Prior treatment with any VEGFR tyrosine kinase inhibitor(such as sunitinib, sorafenib, bevacizumab, imatinib, famitinib, apatinib, regorafenib and other drugs).
* Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy, is planned for the first 4 weeks prior to enrollment or during the study. Radiation radiotherapy (EF-RT) was performed within 4 weeks prior to enrollment.
* A history of other malignancy ≤ 3 years previous
* Known brain metastases.
* The investigator judged that during the follow-up study, the tumor is very likely to invade the important blood vessels and cause fatal hemorrhage, or the formation of tumor thrombosis with large veins (iliac vessels, inferior vena cava, pulmonary veins, superior vena cava);
* The investigator judged that the presence of distinct pulmonary cavitary or necrotic tumors;
* Serosal effusion with clinical symptoms requiring surgical management (including hydrothorax and ascites pericardial effusion)
* with any severe and/or uncontrolled disease, including:1)Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg, despite optimal drug treatment).2)Arrhythmias with grade II and above myocardial ischemia or myocardial infarction, poor control (including corrected QT interval(QTc) men ≥ 450 ms, women ≥ 470 ms) and ≥ 2 congestive heart failure (New York Heart Association ( NYHA) rating).3)Poor control of diabetes (fasting blood glucose > 10mmol / L).4)Active or uncontrolled serious infection (≥ Common Terminology Criteria for Adverse Event(CTC AE) grade 2 infection);5)Patients with active hepatitis B or hepatitis C (hepatitis B: HBsAg-positive and hepatitis B virus(HBV) DNA ≥ 500 IU/mL; hepatitis C: hepatitis C virus(HCV) RNA-positive and abnormal liver function), or active infection requiring antimicrobial treatment (eg Treated with antibacterial drugs, antiviral drugs, antifungal drugs);6)renal insufficiency: urine routine indicates urinary protein ≥ ++, or confirmed 24-hour urine protein ≥ 1.0 g;7)Patients with seizures and need treatment
* Abnormal coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or activated partial thromboplastin time(APTT) > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy.
* Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin.
* significant coughing blood in the 2 months before enrollment, or daily hemoptysis of 2.5ml or more.
* history of psychotropic substance abuse who are unable to quit or have a mental disorder.
* Tendencies of hereditary or acquired hemorrhagic and thrombotic (such as hemophilia patients, coagulopathy, thrombocytopenia, hypersplenism, etc.)
* Any major unhealed wound, ulcer, or fracture occurred in a patient who had undergone major surgery or trauma within 4 weeks and/or had any bleeding or bleeding episodes which the degree is bigger than CTCAE 3 grade within 4 weeks prior to enrollment.
* Active period digestive ulcers.
* Cavity sinus or perforation occurred within 6 months.
* Participated in other anti-tumor clinical trials within 4 weeks.
* Received a potent CYP3A4 inhibitor (such as ketoconazole, itraconazole, erythromycin, and clarithromycin) within 7 days, or received a potent CYP3A4 inducer within 12 days prior to the study (eg. catarrh Treatment with imipramine, rifampicin and phenobarbital).
* Allergic reactions, hypersensitivity reactions or intolerance to anlotinib hydrochloride or its excipients.
* Pregnancy or lactation.
* The investigator believes that there are any conditions that may damage the subject or result in the subject not being able to meet or perform the research request.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Progress free survival | Until Progressive Disease(PD) or death(up to 24 months)
  Progress free survival (PFS) defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.

SECONDARY OUTCOMES:
Overall Survival | From randomization until death (up to 24 months)
  Overall Survival (OS) is defined as the time until death due to any cause.
Objective Response Rate | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective Response Rate (ORR) is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Safety(Number of Participants with Adverse Events and Clinical laboratory numerical evaluation as a Measure of Safety) | Each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Number of Participants with Adverse Events and Clinical laboratory numerical evaluation as a Measure of Safety.

CONTACTS AND LOCATIONS:
Overall Officials: Li Shenglong, master, Principal Investigator — Project sponsor of Liaoning Province Tumor Hospital
Locations (1):
- Liaoning Province Tumor Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chawla SP, Papai Z, Mukhametshina G, Sankhala K, Vasylyev L, Fedenko A, Khamly K, Ganjoo K, Nagarkar R, Wieland S, Levitt DJ. First-Line Aldoxorubicin vs Doxorubicin in Metastatic or Locally Advanced Unresectable Soft-Tissue Sarcoma: A Phase 2b Randomized Clinical Trial. JAMA Oncol. 2015 Dec;1(9):1272-80. doi: 10.1001/jamaoncol.2015.3101. PMID 26378637
- [Result] Spannuth WA, Sood AK, Coleman RL. Angiogenesis as a strategic target for ovarian cancer therapy. Nat Clin Pract Oncol. 2008 Apr;5(4):194-204. doi: 10.1038/ncponc1051. Epub 2008 Feb 12. PMID 18268546